CLINICAL TRIAL: NCT07125573
Title: The Effect of Esketamine Combined With Dexmedetomidine on Postoperative Recovery Quality in Patients Undergoing Thoracoscopic Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Jinqiao Qian, professor, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (2025) Ethical Review L No. 81
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Esketamine Plus Dexmedetomidine Affect Postoperative Quality; Thoracoscopy; Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline solution + dexmedetomidine group (Placebo Comparator): Administer 0.5 ug/kg of dexmedetomidine 10 minutes before surgery, and maintain at 0.4 ug/kg/h after intubation until 30 minutes before the end of surgery,Administer saline solution one minute after induction of anesthesia and continue until 30 minutes before the end of surgery.
  Interventions: Drug: Saline Solution (NaCl 0,9%)
- Low-dose esketamine + dexmedetomidine group (Experimental): Administer dexmedetomidine 0.5 μg/kg 10 minutes before surgery, maintain at 0.4 μg/kg/h after intubation until 30 minutes before the end of surgery, administer esketamine 0.2 mg/kg 1 minute after induction of anesthesia, maintain at 2 μg/kg/min after intubation until 30 minutes before the end of surgery.
  Interventions: Drug: Low-dose esketamine infusion
- High-dose esketamine + dexmedetomidine group (Experimental): Administer 0.5 ug/kg of dexmedetomidine 10 minutes before surgery, and maintain at 0.4 ug/kg/h after intubation until 30 minutes before the end of surgery, Administer 0.2 mg/kg of esketamine 1 minute after induction of anesthesia, and maintain at 4 μg/kg/min after intubation until 30 minutes before the end of surgery.
  Interventions: Drug: High-dose esketamine infusion

INTERVENTIONS:
Drug: Saline Solution (NaCl 0,9%) — Administer 0.5 ug/kg of dexmedetomidine 10 minutes before surgery, and maintain at 0.4 ug/kg/h after intubation until 30 minutes before the end of surgery,Administer saline solution one minute after induction of anesthesia and continue until 30 minutes before the end of surgery.
  Arms: Saline solution + dexmedetomidine group
Drug: Low-dose esketamine infusion — Administer 0.5 ug/kg of dexmedetomidine 10 minutes before surgery, and maintain at 0.4 ug/kg/h after intubation until 30 minutes before the end of surgery, administer esketamine 0.2 mg/kg 1 minute after induction of anesthesia, maintain at 2 μg/kg/min after intubation until 30 minutes before the end of surgery.
  Arms: Low-dose esketamine + dexmedetomidine group
Drug: High-dose esketamine infusion — Administer 0.5 ug/kg of dexmedetomidine 10 minutes before surgery, and maintain at 0.4 ug/kg/h after intubation until 30 minutes before the end of surgery, Administer 0.2 mg/kg of esketamine 1 minute after induction of anesthesia, and maintain at 4 μg/kg/min after intubation until 30 minutes before the end of surgery.
  Arms: High-dose esketamine + dexmedetomidine group

SUMMARY:
Brief Summary：Video-assisted thoracoscopic surgery (VATS) has a wide range of applications, including the diagnosis and treatment of lung cancer, and has gradually replaced traditional open thoracotomy. VATS must routinely employ single-lung ventilation techniques. During single-lung ventilation, mechanical injury, lung collapse, imbalance in the ventilation-perfusion ratio, ischemia-reperfusion, and other pathological physiological changes may occur, leading to the release of a large number of inflammatory factors, triggering local and systemic inflammatory responses,increasing the incidence of postoperative complications, and affecting patient outcomes. Additionally, most patients undergoing thoracoscopic surgery experience acute postoperative pain. If acute postoperative pain is not adequately controlled, it may progress to chronic pain, affecting the quality of postoperative recovery. Currently, opioid medications are the primary drugs used to treat moderate to severe postoperative pain. However, adverse events associated with opioid medications may also affect the quality of postoperative recovery.The use of multimodal analgesia for postoperative pain management can control pain and reduce the need for opioid medications.

Esketamine, a newly marketed intravenous anesthetic in China in recent years, is the dextrorotatory isomer of ketamine, and acts as a non-competitive antagonist of the N-methyl-D-aspartate (NMDA) receptor. Compared to ketamine, esketamine has higher potency, faster recovery time, and fewer adverse effects. Some clinical studies have shown that administration of esketamine reduces the intensity of postoperative pain and decreases the need for postoperative analgesics. Research has found that esketamine reduces the consumption of opioid medications and hyperalgesia postoperatively. Additionally, studies have shown that esketamine administration improves recovery quality by alleviating postoperative pain. Dexmedetomidine (DEX) is a selectiveα2 adrenergic receptor agonist with sedative and analgesic effects. Studies have shown that dexmedetomidine effectively reduces surgical inflammation, oxidative stress, and postoperative pain, thereby promoting postoperative recovery in surgical patients without increasing the risk of adverse reactions or complications. A meta-analysis indicated that dexmedetomidine administration alleviates postoperative pain and reduces postoperative nausea and vomiting (PONV). Current evidence suggests that the use of dexmedetomidine improves postoperative recovery quality. However, the effects of esketamine combined with dexmedetomidine on postoperative recovery quality in patients undergoing thoracoscopic surgery have not been reported. This study aims to investigate whether the combined administration of esketamine and dexmedetomidine can further improve postoperative recovery quality in patients undergoing thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. BMI 18-30 kg/m2;
3. ASA classification I-III;
4. Patients undergoing thoracoscopic surgery;
5. No contraindications to the study drug;
6. Ability to express, communicate, and understand normally;
7. Both the patient and their family members agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Patients with poorly controlled or untreated hypertension;
2. Patients with untreated hyperthyroidism;
3. Patients with mental illness, cognitive impairment, or language barriers that prevent communication;
4. Patients with severe cardiopulmonary, hepatic, or renal dysfunction;
5. Patients with increased intracranial pressure;
6. Patients with a history of allergic reactions to any of the drugs used in the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Record the QoR-15 scale scores for three groups of patients before surgery, on the first day after surgery, and on the third day after surgery. | Record the QoR-15 scale scores for three groups of patients before surgery, on the first day after surgery, and on the third day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

DOCUMENTS (2):
  • Study Protocol (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT07125573/Prot_000.pdf
  • Informed Consent Form (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT07125573/ICF_001.pdf